CLINICAL TRIAL: NCT05401058
Title: Low-dose Droperidol for Prevention of Postoperative Delirium in Elderly Patients After Non-cardiac Surgery: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Low-dose Droperidol for Prevention of Postoperative Delirium in Elderly Patients After Non-cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DECPOD-DP
Record Dates: First submitted 2022-05-23; First posted 2022-06-02 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Digestive System Disease; Urologic Diseases; Gynecological Disease; Orthopedic Surgery
Keywords: non-cardiac surgery; Droperidol; postoperative delirium; elderly patients
MeSH Terms: conditions — Digestive System Diseases; Urologic Diseases; Genital Diseases, Female; Emergence Delirium | interventions — Droperidol; Fumigant 93; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Droperidol 1.25mg/0.5ml
  Interventions: Drug: Droperidol Injection
- Placebo group (Placebo Comparator): Normal saline 0.5ml
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Droperidol Injection — About 30min before the end of operation, Droperidol 1.25mg/0.5ml will be administered by intravenous injection.
  Other Names: D
  Arms: Experimental group
Drug: Saline — About 30min before the end of operation, Normal saline 0.5ml will be administered by intravenous injection.
  Other Names: S
  Arms: Placebo group

SUMMARY:
The aim of this multicenter, prospective, randomized, double-blind and large sample study is to explore the preventive effect of low-dose droperidol on POD in elderly patients after non-cardiac surgery, providing new approach for reducing the incidence of POD and improving the prognosis and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age≥65 years
* American Society of Anesthesiologists (ASA): I-III
* Planning to undergo elective non-cardiac surgery under general anesthesia with endotracheal intubation, including digestive, orthopedic, urologic and gynecological surgery
* Estimated operation time more than 2 hours
* Not expected to be admitted to ICU postoperatively
* Proficient in Chinese
* Informed consent

Exclusion Criteria:

* Morbid obesity with BMI >35 kg/m2;
* History of psychological and neurological diseases, such as depression, schizophrenia, epilepsy, severe central nervous system depression, Parkinson's disease, Alzheimer's disease, myasthenia gravis, basal ganglia disease, etc;
* Corrected QT (QTc) of electrocardiogram> 500ms;
* Preoperative liver insufficiency (Child Pugh grade C);
* End-stage renal disease requiring dialysis;
* Severe heart failure [Metablic equivalent (METs)<4];
* Allergic to droperidol;
* Inability to communicate due to coma or dementia in preoperative period;
* Preoperative delirium, assessed by 3D-CAM;
* More than three standard alcoholic drinks per day (≈10 g alcohol , equivalent to 50 g of strong Chinese spirits);
* Participating in conflicting clinical trials;
* Expected to have an additional operation within 7 days after the index operation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2968 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium within 7 days after operation | 7 days after operation
  Incidence of delirium within 7 days after operation

SECONDARY OUTCOMES:
Severity of delirium | From the end of operation to 7 days after opertation
  Severity of Postoperative delirium
Delirium-free days | From the end of operation to 7 days after opertation
  Delirium-free days
Postoperative hospital duration | From end of operation to discharge, an average of 1 week
  Postoperative hospital duration
cognitive function at 30 days and 6 months | 30 days and 6 months after surgery
  cognitive function at 30 days and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, MD,PHD, Principal Investigator — Renji Hospital, Shanghai Jiaotong University, School of Medcine
Locations (6):
- China (6):
  - The first Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Henan Provincial People Hospital, Zhengzhou, Henan
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Pudong, Shanghai Municipality
  - Second hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Sichuan Academy of Medical Sciences - Sichuan Provincial People's Hospital (SAMSPH), Chengdu, Sichuan
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing